CLINICAL TRIAL: NCT02944370
Title: PlayFit Pilot: Encouraging Social Physical Play in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine, Division Chief of Population Health, Research and Development, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4785
Record Dates: First submitted 2016-10-17; First posted 2016-10-25 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PlayFit, Modified exercise games (Experimental): Subjects will participate in three 60 minute game sessions each week for 12 weeks. During each game session, subjects will be divided randomly into two teams to play a modified game. Research staff will review the instructions of the game and if needed, modify the game rules during play to enhance the experience (ie. keep it fun, keep it to moderate intensity level). The length of play session between breaks increases each week.
  Interventions: Behavioral: PlayFit - modified exercise games

INTERVENTIONS:
Behavioral: PlayFit - modified exercise games — Play modified games with other adults three times a week for 12 weeks. Complete a brief survey on the games played and program satisfaction.

SUMMARY:
The investigator is pilot testing the feasibility and impact of a low-cost intervention that uses existing gymnasiums, and therefore has the potential to be replicated across the United States. The intervention, PlayFit, is designed for adults aged 21-50. PlayFit has five key components, intended to overcome the major barriers to physical activity. First, it will assist people in finding others to play with, using the Pick-Up model of designating times to play and making those times known in the community. Second, it will overcome a lack of confidence in physical activity by including games of lower intensity for relatively unfit adults, then building up to moderate and vigorous games. Third, it will require team members of varying ages and genders to encourage intergenerational play. Fourth, it will use modified equipment (e.g., softer, lighter balls) and smaller game space to require less running, so that even relatively unfit people can feel confident participating. Fifth, it will be designed to be led by community volunteers, which will increase its disseminability.

AIM - Understand the optimum design for PlayFit. To meet this aim, the investigators will come up with a list of games to play and pilot the games at a gymnasium. The investigators will observe the participants playing the games and have them complete a brief survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-50
* Fluently read and speak English
* Current member of Hershey Medical Center's University Fitness Center OR willing to become a member
* Currently exercises < 150 minutes per week

Exclusion Criteria:

* Has been told by a doctor they a heart condition and should only do exercise recommended by a doctor
* Currently pregnant or planning to become pregnant in the next 6 months
* Planning to move out of the area in the next 6 months
* Has pain in chest, neck, jaw, or arms at rest, during daily activities of living
* Has experienced a forceful or rapid heart rate
* Has experience unreasonable breathlessness
* Has experienced dizziness fainting or blackouts
* Has experienced ankle swelling
* Has burning or cramping sensation in lower legs when walking short distances
* Has been told by a health professional not to exercise OR exercise only when supervised by a professional
* Has been diagnosed with diabetes
* Has been told by a doctor, nurse or health professional that they have (1) Weak or failing kidneys, (2) A heart attack/ myocardial infarction, (3) Angina or coronary heart disease, (4) A stroke, or (5) Any other kind of heart condition or heart disease - e.g. heart valve problem/aortic regurgitation (do not include heart murmur)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Compare exercise intensity, METS (Metabolic Equivalent Task) | 12 weeks
  METS will be measured during each exercise session using an accelerometer (ActiGraph GT3X).

SECONDARY OUTCOMES:
Self-reported weight | 12 weeks
  Self-reported weight will be captured by a research assistant at baseline and follow up (12 week) visits.
Self-reported height | 12 weeks
  Self-reported height will be captured by a research assistant at baseline and follow up (12 week) visits.
Gender | 12 weeks
  Participants will be asked if they are male or female.
Self-reported chronic conditions | 12 weeks
  Participants will be asked 4 questions on which chronic conditions (if any) they may have.
Ethnicity | 12 weeks
  Participants will be asked what their ethnicity is.
Race | 12 weeks
  Participants will be asked what their race is.
Education Level | 12 weeks
  Participants will be asked 1 question on education level.
Employment Status | 12 weeks
  Participants will be asked 1 question on employment status.
Tobacco Use | 12 weeks
  Participants will be asked 1 question on tobacco use.
National Health Interview Survey | 12 weeks
  Participants will be asked 2 questions from this survey on how difficult it is to walk and carry an item.
General Self Rated Health | 12 weeks
  Participants will be asked 1 question on their overall health.
Three Item Loneliness Scale | 12 weeks
  Participants will be asked 3 questions on feelings of being lonely.
Patient Reported Outcomes (PROMIS) - Anxiety | 12 weeks
  Participants will be asked questions 4 questions on anxiety.
Patient Reported Outcomes (PROMIS) - Depression | 12 weeks
  Participants will be asked 4 questions on Depression.
Patient Reported Outcomes (PROMIS) - Physical Function | 12 weeks
  Participants will be asked 4 questions on physical function.
Sport playing status | 12 weeks
  Participants will be asked 2 questions on playing sports previously.
Program Intensity Survey | 12 weeks
  Participants will be asked 2 questions after each game session on how physically and technically hard the game was.
Program Satisfaction Survey | 12 weeks
  Participants will be asked 2 questions after each game session on what they did and did not like about the game.
Net Promoter Score | 12 weeks
  Participants will be asked 1 question on how likely they would recommend the day's activity/game to a friend or family member.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States